CLINICAL TRIAL: NCT02042664
Title: Effect of GLP-1 Receptor (GLP-1R) Agonists on Cardiac Function and on Epicardial Adipose Tissue (EAT) Volume and on Myocardial TG Content in Obese Diabetics
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010 -022792-57; 2010-14 (Other: AP HM)
Record Dates: First submitted 2013-09-11; First posted 2014-01-23 (Estimated); Last update posted 2015-08-31 (Estimated); Status verified 2015-08

CONDITIONS: Obesity; Diabetes
MeSH Terms: conditions — Obesity; Diabetes Mellitus | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- treatment BYETTA (Experimental)
  Interventions: Drug: BYETTA treatment
- metformine (Active Comparator)
  Interventions: Drug: Metformine

INTERVENTIONS:
Drug: BYETTA treatment
  Arms: treatment BYETTA
Drug: Metformine
  Arms: metformine

SUMMARY:
Glucagon-like peptide-1 (GLP-1) receptor agonist are new treatment of type 2 diabetes, they lower blood glucose level (by enhancement of glucose-dependent insulin secretion and suppression of excess glucagon secretion) and reduce weight by inducing satiety and slowing of gastric emptying. Beneficial effects of GLP-1 and GLP-1 receptor (GLP-1R) agonists on cardiovascular function have been suggested. They improve biomarkers of CV risk, decrease systolic blood pressure, improve endothelial function and have beneficial effects on myocardium. Nevertheless, few studies have analysed the effect of GLP1 treatment on myocardial function in type 2 obese diabetic.

Myocardial steatosis is an independent predictor of diastolic dysfunction in type 2 diabetes mellitus. It was recently shown that 16 weeks of caloric restriction in obese patients with diabetes decrease myocardial triglyceride content and improve myocardial function (cardiac output, normalized stroke volume, LV mass and normalized end diastolic volume), and diastolic function. However, no study has evaluated the impact of Glucagon-like peptide-1 (GLP-1) receptor agonist in obese diabetics on myocardial TG content.

Recent studies have suggested that increased epicardial adipose tissue (EAT) could be an important risk factor for cardiac diseases. We and others have already evidenced a correlation between the volume of epicardial adipose tissue and the presence or the severity of coronaropathy. The impact of weight loss on the volume of EAT or the characteristics of EAT is mostly unknown.

ELIGIBILITY:
Inclusion Criteria:

* - Patients with type 2 diabetes according to WHO criteria
* Age> 18 years
* BMI ≥ 30 kg/m2
* HbA1c> 7% and <10%
* Processing by ADO (Metformin and Glimepiride)
* Effective contraception (for women)
* Signed informed consent by the patient before inclusion in the protocol

Exclusion Criteria:

* Ongoing pregnancy or become pregnant within six months of the study protocol
* Breastfeeding
* Recent weight loss (> 5% of total weight)
* Treatments changing the distribution of adipose tissue as corticosteroids or glitazones
* Acute coronary syndrome or unstable angina during the last three months
* Contraindications to cardiac MRI (mechanical heart valve, pacemaker, metallic intraocular foreign body, claustrophobia)
* Contraindication to cold test: Raynaud's syndrome
* Contraindication to exenatide:

  * Neoplasia active or untreated or in remission for less than 5 years (except for basal cell carcinoma or in situ cervical or prostate)
  * Contraindication to ADO (depending on specific product) in combination with exenatide.
  * History of kidney transplant or dialysis or plasmatique creatinine> 1.5 mg / dL for men and> 1.2 mg / dL for women
  * Digestive diseases, including gastroparesis
  * plasma triglycerides> 1000 mg / dL
  * History of pancreatitis confirmed biologically
  * contraindication or hypersensitivity to Exenatide or one of its social coverage composantsAbsence

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2011-01; Primary Completion 2015-01 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
intracardiac triglyceride | 3 years
  Cardiac MRI

CONTACTS AND LOCATIONS:
Overall Officials: LOIC modoloni, Study Director — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France

REFERENCES:
- [Derived] Soghomonian A, Dutour A, Kachenoura N, Thuny F, Lasbleiz A, Ancel P, Cristofari R, Jouve E, Simeoni U, Kober F, Bernard M, Gaborit B. Is increased myocardial triglyceride content associated with early changes in left ventricular function? A 1H-MRS and MRI strain study. Front Endocrinol (Lausanne). 2023 Jun 22;14:1181452. doi: 10.3389/fendo.2023.1181452. eCollection 2023. PMID 37424866